CLINICAL TRIAL: NCT04715100
Title: Relationship of Pain and Joint Status With the Perception of Psychosocial Factors in Patients With Hemophilic Arthropathy: A Multicenter Observational Study
Brief Title: Pain and Joint Status With Psychosocial Factors in Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Other Study IDs: He-Perception
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia Arthropathy
Keywords: Hemophilic arthropathy; Educational intervention; Joint pain; Quality of life; Anxiety; Stress
MeSH Terms: conditions — Arthralgia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: The inclusion criteria to participate in the present study are patients: with a diagnosis of hemophilia A and B; adults; and on a prophylactic or on-demand treatment regimen with FVIII / FIX concentrates.
  For their part, patients with: neurological or cognitive alterations that impede understanding of the questionnaires will be excluded from the study; Dependent patients who require help from a third person to get around; patients who have developed a hemarthros in the 4 weeks prior to the study; and those who have not signed the informed consent document.
  For inclusion in the study, patients will continue to be administered the dose of FVIII / FIX concentrates, following the guidelines of the medical criteria established by their reference hematologist. Throughout this study, the medical criteria for drug treatment, the dosage, and the replacement treatment periods will not be changed.
  Interventions: Other: Observational group

INTERVENTIONS:
Other: Observational group — The study dependent variables will be: pain (vas scale), joint status (Hemophilia Joint Health Score), perception of quality of life (SF-36 questionnaire), list of roles (Oakley questionnaire), performance of basic activities of daily life (Barthel index) and the performance of instrumental activities of daily living (Lawton and Brody scale).

SUMMARY:
Background. The recurrence of hemarthrosis in patients with congenital coagulopathies favors the development of a progressive, degenerative intra-articular lesion (hemophilic arthropathy) that mainly affects the knees, ankles and elbows. Disability and functional limitations are characteristic sequelae of these patients from an early age.

Objective. To assess the joint status, the perception of quality of life, the performance of roles and the performance of daily life activities, in patients with hemophilic arthropathy.

Study design. Observational, multicenter study. Method. 70 patients with hemophilia A and B will be included in this study. Patients will be recruited from 4 centers in different regions of Spain. The dependent variables will be: pain (measured with the Visual Analogue Scale), joint status (Hemophilia Joint Health Score), perception of quality of life (SF-36 questionnaire), list of roles, performance of daily life activities (Barthel scale), performing the instrumental activities of daily life (Lawton and Brody scale). The evolution of the variables will be analyzed using parametric (t-student or ANOVA) or non-parametric (Wilcoxon or Friedman) tests. A correlation analysis will be carried out between the dependent and independent variables, as well as a linear regression analysis between the observed determining variables.

Expected results. The aim is to observe the relationship of pain and joint status in patients with hemophilic arthropathy, with their perception of quality of life, the development of the roles they play and the performance of basic and instrumental activities of daily living.

DETAILED DESCRIPTION:
Main objective: To analyze the relationship of pain and joint status with psychosocial and functional variables in adult patients with hemophilic arthropathy.

Secondary objectives: i) To detect the relationship between joint damage in psychosocial disorders in patients with hemophilia; ii) Evaluate the performance and perception of roles with the clinical situation of patients with hemophilic arthropathy; iii) Identify the factors that influence the performance of basic and instrumental activities of daily living in adult patients with hemophilia; iv) Observe changes in the perception of quality of life, performance of roles and activities of daily life based on the clinical and sociodemographic characteristics of patients with hemophilia.

Patients who meet the selection criteria will be summoned to a meeting where the principal investigator will present, orally and in writing, the characteristics of the investigator, the intended objectives and the risks of the intervention. At said meeting, the following documentation will be provided: patient information document and informed consent document for patients.

After obtaining the informed consent of the patients, the evaluations will be carried out in the dependencies of the locations included in the study. Six dependent variables will be measured: pain, joint condition, perception of quality of life, list of roles, performance of basic activities of daily life, and performance of instrumental activities of daily life.

All joint state evaluations will be performed by the same physiotherapist, blinded to the objectives of the study. The evaluation of the questionnaires will be analyzed by another evaluator, blinded to the objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B
* Patients of legal age
* Patients on prophylactic or on demand treatment with clotting factor concentrates.

Exclusion Criteria:

* Patients with neurological or cognitive disorders that impede the understanding of the questionnaires
* Dependent patients who require help from a third person to get around
* Patients who have developed a hemarthros in the 4 weeks prior to the study.
* Patients who have not signed the informed consent document.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia attending in hemophilia Associations into Spanish Federation of Hemophilia (Fedhemo).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess the perception of joint pain with numerical scale of pain | Screening visit
  Measurement with numerical scale of pain. The patient must assign pain to a numerical value between two extreme points (0 to 10). Although the subject is asked to use numerical values to indicate the level of pain, the use of keywords, as well as previous instructions, are necessary if we expect the patient to conceptualize their pain in numerical terms. The scale is discrete, not continuous, but to perform statistical analyzes, equal intervals can be assumed between categories (score 0-10; higher scores mean a worse joint pain).
Assess the joint status with Hemophilia Joint Health Score | Screening visit
  Measurement the joint status with the instrument: Haemophilia Joint Health Score (score 0-120; higher scores mean a worse joint status).

SECONDARY OUTCOMES:
Assess the perception of quality of life with the questtionaire Short Form 36 Health Survey | Screening visit
  Measurement with Short Form 36 Health Survey [SF-36]. This health questionnaire is one of the most widely used, validated and translated instruments in the field of measuring the quality of life related to health. The SF-36 health questionnaire is a generic instrument consisting of 36 questions, which provides a profile of the health status and is applicable to both patients and the healthy population. The questionnaire covers 8 dimensions: physical functioning, physical role, corporal pain, general health, vitality, social functioning, emotional role and mental health of the patient. (score 0-100; higher scores mean a better outcome).
Assess the list of roles with Oakley scale | Screening visit
  It will be measured with Oakley et al (1985). The list is divided into 2 parts: the first assesses the roles that have served the most to organize the individual's daily life and the second identifies the degree to which the individual values each role. The list presents 10 roles: student, worker, caregiver, homeowner, friend, family member, religious participant, hobbyist, and participant in organizations. The list aims to identify the roles that organize the individual's daily life, for this reason the definition of each role refers to the frequency of performance. (score 0-60; higher scores mean a better outcome).
Assess the carrying out activities of daily living | Screening visit
  It will be measured with the Barthel index. This scale measures the capacity of the person to carry out ten basic activities of daily life, obtaining a quantitative estimate of the degree of dependence of the subject. This instrument assesses each of the corresponding activities and, depending on your ability to perform it, scores with 0, 5 or 10 points (up to 15 for certain activities). (score 0-100; higher scores mean a better outcome).
Assess the instrumental activities of daily living | Screening visit
  It will be evaluated with the Lawton and Brody scale. This questionnaire measures the degree of independence that the patient maintains. It is made up of eight items with various response alternatives that together evaluate the ability to carry them out autonomously. The answer options score 1 (the person performs them independently) or 0 (dependent). (score 0-8; higher scores mean a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seoane-Martin ME, Cuesta-Barriuso R, Rodriguez-Martinez MC. Performance of instrumental activities of daily living in patients with haemophilic arthropathy. A cross-sectional cohort study. Haemophilia. 2024 Nov;30(6):1406-1413. doi: 10.1111/hae.15114. Epub 2024 Oct 24. PMID 39447049